CLINICAL TRIAL: NCT04204356
Title: The Effect of Speech and Language Therapy With and Without Transcranial Direct-current Stimulation on Discourse Production in People With Post-stroke Aphasia: a Pilot Randomised Controlled Trial
Brief Title: The Effect of Non-invasive Brain Stimulation on Language Production in Post-stroke Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HR-19/20-12921
Record Dates: First submitted 2019-12-13; First posted 2019-12-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Aphasia; Stroke; Language Disorders
MeSH Terms: conditions — Aphasia; Stroke; Language Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS group (Experimental): Participants randomly allocated to this group using a random number generator will receive a once weekly, 6-week block of language treatment with active tDCS.
  Interventions: Behavioral: Language treatment for improving discourse production; Device: Transcranial direct-current stimulation (tDCS)
- Sham group (Sham Comparator): Participants randomly allocated to this group using a random number generator will receive a once weekly, 6-week block of language treatment without active tDCS (sham)
  Interventions: Behavioral: Language treatment for improving discourse production

INTERVENTIONS:
Behavioral: Language treatment for improving discourse production — All participants will receive a 6-week block of language treatment for improving verb retrieval in discourse production by a professional speech and language therapist. The treatment goals for this block of treatment are to 1) improve verb retrieval and language quantity and complexity in discourse production 2) improve functional communication skills and; 3) improve quality of life and psychological state in people with post-stroke chronic aphasia.
Device: Transcranial direct-current stimulation (tDCS) — Transcranial direct-current stimulation is a non-invasive brain stimulation method that can modify spontaneous cortical activity in targeted brain regions. Anodal tDCS delivered through a positively charged electrode has been found to increase cortical excitability in a targeted brain region. The use of tDCS as an adjunct to speech and language therapy has been found to improve aphasia treatment effects in post stroke patient populations.
  Arms: tDCS group

SUMMARY:
Aphasia is a language impairment caused by brain injury such as stroke that affects the ability to understand and express language, read and write due to damage in the language regions of the brain. Non-invasive brain stimulation (NIBS) techniques like transcranial direct-current stimulation (tDCS) have been found to improve aphasia treatment effects in post stroke patient populations such as improved naming abilities.

However, the effect of tDCS on more functional, higher level language skills such as discourse production (i.e. story telling, giving instructions) has yet to be understood.Therefore the aim of this study is to determine the potential effectiveness of tDCS as an adjunct to speech and language therapy (SLT) to improve discourse speech production in people with post-stroke aphasia. It is hypothesised that SLT combined with tDCS will result in greater improvements in discourse language production compared to SLT on its own.

ELIGIBILITY:
Inclusion Criteria:

* aphasia caused by a single stroke
* at least 6 months post stroke
* at least 18 years old
* competent English speaker prior to stroke
* right handed prior to stroke
* normal aided or unaided visual acuity
* willing to participate and to comply with the proposed block of intervention and testing regime.

Exclusion Criteria:

Persons with

* neurological symptoms or history of a neurological event other than their stroke
* contraindications to tDCS including history of epilepsy or seizures and pacemakers
* global/severe aphasia
* cognitive impairment identified by a score less than 20/30 in the Montreal Cognitive Assessment
* left-handed dominance prior to stroke
* visual problems which interfere with persons' ability to access visual materials (i.e. pictures)
* inability to attend sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Verb token total | 30 minutes
  The number of all verb occurrences in a language sample
Verb type total | 30 minutes
  The number of distinct verbs in a sample

SECONDARY OUTCOMES:
Total number of words | 30 minutes
  The total number of words in a language sample
Total number of utterances | 30 minutes
  The total number of utterances in a language sample
Predicate argument structure (PAS) | 30 minutes
  The main verbs and their arguments will be identified in each sentence within a language sample. A PAS complexity score will be calculated using the formula: number of arguments/number of main verbs
Communicative Effectiveness Index (CETI) | 10 minutes
  CETI is a valid and reliable measure of change in functional communication ability in adults with aphasia. This assessment includes 16 everyday situations such as having a one to one conversation and giving yes or no answers appropriately. Participants are asked to rate their ability in each particular communication situation using a rating scale with one end labelled as 'not at all able and the other 'as able as before
Aphasia Impact Questionnaire-21 (AIQ) | 15 minutes
  AIQ is a self-report questionnaire which utilises pictures to enable people with aphasia to communicate their experiences of aphasia. There are 8 questionnaires to select from with scales that vary in relation to gender and race. Pictorial responses can be translated into numerical scores, and then documented on a summary score sheet. The questionnaire has three sections; communication, participation and well-being/emotional state. The first section looks at activities which are commonly difficult for people with aphasia such as talking and understanding. The participation section looks at how communication difficulties arising from aphasia impact the person's ability to complete tasks in everyday life such as shopping and work. The last section looks at the emotional effect of aphasia.
Hospital Anxiety and Depression Scale (HADS) | 10 minutes
  HADS is a 14-item scale which assesses non-somatic anxiety and depression symptoms. Scores range from 0 to 21 for each sub-scale with a score ≥8 proposed for the identification of caseness, for both depression and anxiety.
Montreal Cognitive Assessment (MoCA) | 15 minutes
  The MoCA is a brief and easy to administer cognitive assessment. Different aspects of cognition such as memory, executive function, language, visual-spatial ability and orientation are assessed. Scores range from 0-30, where the recommended cut-off score for identifying multi-domain cognitive impairment in persons with chronic stroke is 20/30.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All information collected will be kept confidential and stored anonymously on password protected computers used only by research staff who are part of the study. Data will be stored securely in accordance with the Data Protection Act (1998) and the General Data Protection Regulations (May 2018). Stored, anonymised data may be used for future medical and health-related studies. Anonymised data will be retained for 10 years.

REFERENCES:
- [Background] Lambon Ralph MA, Snell C, Fillingham JK, Conroy P, Sage K. Predicting the outcome of anomia therapy for people with aphasia post CVA: both language and cognitive status are key predictors. Neuropsychol Rehabil. 2010 Apr;20(2):289-305. doi: 10.1080/09602010903237875. Epub 2010 Jan 1. PMID 20077315
- [Background] Coelho CA, Liles BZ, Duffy RJ. Contextual influences on narrative discourse in normal young adults. J Psycholinguist Res. 1990 Nov;19(6):405-20. doi: 10.1007/BF01068887. PMID 2286935
- [Background] Brady MC, Kelly H, Godwin J, Enderby P. Speech and language therapy for aphasia following stroke. Cochrane Database Syst Rev. 2012 May 16;(5):CD000425. doi: 10.1002/14651858.CD000425.pub3. PMID 22592672
- [Background] Holland R, Leff AP, Josephs O, Galea JM, Desikan M, Price CJ, Rothwell JC, Crinion J. Speech facilitation by left inferior frontal cortex stimulation. Curr Biol. 2011 Aug 23;21(16):1403-7. doi: 10.1016/j.cub.2011.07.021. Epub 2011 Aug 4. PMID 21820308
- [Background] Marangolo P, Fiori V, Calpagnano MA, Campana S, Razzano C, Caltagirone C, Marini A. tDCS over the left inferior frontal cortex improves speech production in aphasia. Front Hum Neurosci. 2013 Sep 6;7:539. doi: 10.3389/fnhum.2013.00539. eCollection 2013. PMID 24046740
- [Background] Monti A, Ferrucci R, Fumagalli M, Mameli F, Cogiamanian F, Ardolino G, Priori A. Transcranial direct current stimulation (tDCS) and language. J Neurol Neurosurg Psychiatry. 2013 Aug;84(8):832-42. doi: 10.1136/jnnp-2012-302825. Epub 2012 Nov 8. PMID 23138766
- [Background] Baker JM, Rorden C, Fridriksson J. Using transcranial direct-current stimulation to treat stroke patients with aphasia. Stroke. 2010 Jun;41(6):1229-36. doi: 10.1161/STROKEAHA.109.576785. Epub 2010 Apr 15. PMID 20395612
- [Background] Carroll C, Guinan N, Kinneen L, Mulheir D, Loughnane H, Joyce O, Higgins E, Boyle E, Mullarney M, Lyons R. Social participation for people with communication disability in coffee shops and restaurants is a human right. Int J Speech Lang Pathol. 2018 Feb;20(1):59-62. doi: 10.1080/17549507.2018.1397748. Epub 2017 Dec 1. PMID 29192805
- [Background] Marangolo P, Fiori V, Campana S, Calpagnano MA, Razzano C, Caltagirone C, Marini A. Something to talk about: enhancement of linguistic cohesion through tdCS in chronic non fluent aphasia. Neuropsychologia. 2014 Jan;53:246-56. doi: 10.1016/j.neuropsychologia.2013.12.003. Epub 2013 Dec 11. PMID 24333381
- [Background] Brady MC, Kelly H, Godwin J, Enderby P, Campbell P. Speech and language therapy for aphasia following stroke. Cochrane Database Syst Rev. 2016 Jun 1;2016(6):CD000425. doi: 10.1002/14651858.CD000425.pub4. PMID 27245310
- [Background] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving aphasia in patients with aphasia after stroke. Cochrane Database Syst Rev. 2015 May 1;(5):CD009760. doi: 10.1002/14651858.CD009760.pub3. PMID 25929694
- [Background] Newton C, Kirby P, Bruce C. Getting into shape: the effect of Shape Coding on the spoken language production of two men with chronic aphasia. Aphasiology. 2017;31(12):1459-1481. doi:10.1080/02687038.2017.1306639
- [Background] Pritchard M, Hilari K, Cocks N, Dipper L. Psychometric properties of discourse measures in aphasia: acceptability, reliability, and validity. Int J Lang Commun Disord. 2018 Nov;53(6):1078-1093. doi: 10.1111/1460-6984.12420. Epub 2018 Aug 28. PMID 30155970
- [Background] Lomas J, Pickard L, Bester S, Elbard H, Finlayson A, Zoghaib C. The communicative effectiveness index: development and psychometric evaluation of a functional communication measure for adult aphasia. J Speech Hear Disord. 1989 Feb;54(1):113-24. doi: 10.1044/jshd.5401.113. PMID 2464719
- [Background] Swinburn K. Aphasia Impact Questionnaire. Connect Commun Disabil Netw. 2015. http://www.ukconnect.org/professionals/aiq.
- [Background] Chiti G, Pantoni L. Use of Montreal Cognitive Assessment in patients with stroke. Stroke. 2014 Oct;45(10):3135-40. doi: 10.1161/STROKEAHA.114.004590. Epub 2014 Aug 12. No abstract available. PMID 25116881
- [Background] Kang EK, Kim YK, Sohn HM, Cohen LG, Paik NJ. Improved picture naming in aphasia patients treated with cathodal tDCS to inhibit the right Broca's homologue area. Restor Neurol Neurosci. 2011;29(3):141-52. doi: 10.3233/RNN-2011-0587. PMID 21586821
- [Background] Ross LA, McCoy D, Wolk DA, Coslett HB, Olson IR. Improved proper name recall by electrical stimulation of the anterior temporal lobes. Neuropsychologia. 2010 Oct;48(12):3671-4. doi: 10.1016/j.neuropsychologia.2010.07.024. Epub 2010 Jul 24. PMID 20659489